CLINICAL TRIAL: NCT06128772
Title: A Randomized Clinical Trial Utilizing Battlefield Acupuncture to Treat Chronic Pain in Veterans With a History of Substance Use Disorder.
Brief Title: Utilizing Battlefield Acupuncture to Treat Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edith Nourse Rogers Memorial Veterans Hospital (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cathy St. Pierre, Principal Investigator, Edith Nourse Rogers Memorial Veterans Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1765968
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain; Substance Use Disorders
Keywords: Veterans; chronic pain; Substance Use History; Battlefield Acupuncture
MeSH Terms: conditions — Chronic Pain; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (Other): Eight weeks of waitlist control and then 8 weeks of weekly treatment
  Interventions: Other: Battlefield Acupuncture
- Immediate treatment (Other): Eight weeks of weekly treatment and then eight weeks of follow up
  Interventions: Other: Battlefield Acupuncture

INTERVENTIONS:
Other: Battlefield Acupuncture — 5 points of acupuncture treatment in each ear weekly for 8 weeks

SUMMARY:
This research study will evaluate the effectiveness of utilizing Battlefield Acupuncture (BFA) on veterans with with a history of substance use disorder and chronic pain for 8 weeks.

Primary Aim: The primary aim of this study is to evaluate the effectiveness of using BFA to treat chronic pain in veterans with a history of substance use disorder.

Secondary Aim: This study will also evaluate the impact that BFA treatment for pain may have on subjects' stress, mood and sleep patterns over 8 weeks. In addition, each subject will be complete behavioral research tools to measure: depression, anxiety, and substance use at 3 different points in this study.

Hypothesis: The use of BFA on veterans with chronic pain will decrease their pain and substance use and improve their quality of life.

DETAILED DESCRIPTION:
Objective(s): This research study will evaluate the effectiveness of utilizing Battlefield Acupuncture (BFA) on veterans with with a history of substance use disorder and chronic pain for 8 weeks.

Primary Aim: The primary aim of this study is to evaluate the effectiveness of using BFA to treat chronic pain in veterans with a history of substance use disorder.

Secondary Aim: This study will also evaluate the impact that BFA treatment for pain may have on subjects' stress, mood and sleep patterns over 8 weeks. In addition, each subject will be complete behavioral research tools to measure: depression, anxiety, and substance use at 3 different points in this study.

Hypothesis: The use of BFA on veterans with chronic pain will decrease their pain and substance use and improve their quality of life.

2. Research Design: This is a prospective, RCT trial research study recruiting veterans with a history of chronic pain and substance use disorder.

3.3 Study Procedures

1. Sub-Study Participation- N/A.
2. Study A sample of veterans with chronic pain and substance use disorder will be recruited through distribution of flyers, live or virtual presentations, regarding this study.

   Interested veterans will attend an overview/orientation of this study. Recruited subjects will be given an informed consent (IFC) to read and sign. After completion of IFC the initial research packet will be given to complete and return to the research team.

   Once enrolled, each subject will be assigned to a wait list control of 8 weeks or active treatment for 8 weeks.

   Those in active treatment will be given a 15-20 minute appointment treatment time for the duration of 8 weeks.

   At each appointment, the subject will complete the BFA Questionnaire and other measures, prior to BFA treatment. Prior to treatment, the PI will briefly review subjects questionnaires and answer any questions. The PI will then provide the treatment.

   Treatment with BFA will include placing up to 5 BFA tacks in each ear, for a total of 10 per treatment. Each subject will provide a pain score in the following sequence: pre-treatment, after 3 BFA needles are placed in each ear and again, after the last 2 needles are placed.

   Post treatment instructions will be reviewed and PI will answer any questions. At the completion of the clinic, a note will be recorded in each subject's chart.

   All completed questionnaires will be kept in a locked file cabinet in the PI's locked office. Data will be coded and analyzed at a later time.

   There are no other examinations included for this study. A member of the research team will code each visit and transcribe de-identified data into a codebook.

   3. Methodology: This is a RCT design study. A total of 60 subjects will be recruited for this study. The primary study outcome variables are: substance use and pain level- pre and post treatment, stress, mood and usual activity levels, sleep patterns and behavioral factors such as anxiety and depression.

   4. Findings: Pending

   5. Clinical Relationships: This study is conducted to demonstrate whether or not BFA treatment will decrease pain and improve quality of life for veterans with chronic pain and substance use disorder.

   6. Impact/Significance: Pending

ELIGIBILITY:
Inclusion Criteria: Eligibility criteria include:

* they are 18 years or older
* they have a history of substance use disorder,
* history of chronic pain
* availability to participate in the study for 16 weeks.

Exclusion Criteria:

* female veterans who are pregnant.
* history of bleeding disorders or currently on older blood thinning medications that cause excessive bleeding.
* currently being treated for an active infection of the outer ear (relative contraindication). -- currently have a PICC line in their body or are receiving IV antibiotics.
* fear of needles/tacks, and/or
* undiagnosed pain complaint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Acupuncture questionnaire evaluating chronic pain levels | 8 weeks of treatment, 8 weeks of post treatment follow-up
  Chronic pain level questionnaire ( Acupuncture questionnaire consists of X questions regarding pain. Patients select the level of pain from 0-10 ( the higher the number, the higher the pain. The scale range would be = (0-60).

SECONDARY OUTCOMES:
Acupuncture Follow up Questionnaire which also evaluates the impact that BFA treatment for pain may have on subjects' stress, mood and sleep patterns over 8 weeks. | 8 weeks of treatment and 8 weeks of follow up
  weekly evaluation of subjects' stress, mood and sleep patterns over 8 weeks. Each question is followed by the pain scale which is from 0-10 (the higher the number, the more pain the patient is experiencing as it relates to the impact of pain on their sleep, mood, stress level and activity.
PHQ-4 | monthly for 16 weeks
  monthly evaluation of subjects' mood, anxiety level and depression level
Substance Use Questionnaire- | monthly for 16 weeks
  Questionnaire evaluating subjects' lifetime and recent substance(s) use.

CONTACTS AND LOCATIONS:
Locations (1):
- Bedford VA Healthcare System, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No